CLINICAL TRIAL: NCT01624740
Title: Precision Plus™ High-Rate Subperception SCS for the Treatment of Chronic Intractable Pain
Brief Title: High Rate Spinal Cord Stimulation (SCS) for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A7001
Record Dates: First submitted 2012-06-15; First posted 2012-06-21 (Estimated); Results first posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Rate Followed By High Rate (Experimental): The Precision Plus spinal cord stimulation screening trial leads were temporarily implanted by the investigator. Subjects received low rate stimulation (2 Hz) for 3-4 days, followed by high rate stimulation (1200 Hz) for 3-4 days.
  Interventions: Device: Low Rate Stimulation; Device: High Rate Stimulation
- High Rate Followed By Low Rate (Experimental): The Precision Plus spinal cord stimulation screening trial leads were temporarily implanted by the investigator. Subjects received high rate stimulation (1200 Hz) for 3-4 days, followed by low rate stimulation (2 Hz) for 3-4 days.
  Interventions: Device: Low Rate Stimulation; Device: High Rate Stimulation

INTERVENTIONS:
Device: Low Rate Stimulation — Stimulation was given at a rate of 2 Hz.
Device: High Rate Stimulation — Stimulation was given at a rate of 1200 Hz.

SUMMARY:
To determine the effects of varying spinal cord stimulation programming parameters, including stimulation rate, on pain intensity.

DETAILED DESCRIPTION:
This study compared the effects of high-rate subperception stimulation with the effects of low-rate subperception stimulation on pain intensity.

ELIGIBILITY:
Inclusion Criteria:

* Chronic intractable pain of the trunk and/or limbs
* Documented history of trunk and/or limb pain of at least 180 days
* Average back pain intensity of 5 or greater on a 0-10 numerical rating scale during the 7-day period prior to the Screening Visit
* Pass study site's routine psychological/psychiatric evaluation within 180 days of the Trial Lead Insertion Visit
* If taking any medications for chronic pain, must be on a stable prescription during the 14-day period prior to the Trial Lead Insertion Visit and agree to continue on the same prescription throughout study participation
* Subject is willing and able to comply with all protocol-required procedures and assessments/evaluations
* Subject is able to independently read and complete all questionnaires and/or assessments provided in English
* 18 years of age or older when written informed consent is obtained
* Subject signs a valid, Institutional Review Board (IRB)-approved informed consent form (ICF) provided in English

Exclusion Criteria:

* Unable to operate the Precision Plus system
* Primary source of pain is cancer-related, pelvic, visceral, angina, or migraine
* Is a high surgical risk
* Is diabetic
* Is immunocompromised
* Currently on any anticoagulant medications that cannot be discontinued during perioperative period
* Untreated major depression or untreated generalized anxiety disorder
* Diagnosed with somatoform disorder, severe personality disorder, borderline personality disorder
* Diagnosed with any major psychiatric disorder not specifically listed in CE7 or CE8
* Currently diagnosed with cognitive impairment that would limit subject's ability to discern differences in pain severity, complete a pain diary, perform wound care
* Current abuse of alcohol or illicit drugs
* Subject requires Magnetic Resonance Imaging (MRI) while implanted with lead(s).
* Subject is participating (or intends to participate) in another drug or device clinical trial that may influence the data that will be collected for this study
* Subject has previously undergone a spinal cord stimulation trial or is already implanted with an active implantable device(s) to treat their pain (Implantable Pulse Generators (IPGs), implantable drug pump, etc.) or pacemaker or implantable cardiac defibrillator
* Patient is a woman who is not using adequate contraception, is pregnant or breastfeeding or intends to become pregnant during the course of the study (a urine pregnancy test must be performed within 28 days prior to the Trial Lead Insertion Visit in women of child-bearing potential and the test result documented)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omid Khodai, OD, Study Director — Boston Scientific Corporation
Locations (1):
- Coastal Pain Spinal Diagnostic, Carlsbad, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 20 subjects enrolled (11 to receive low rate stimulation first, 9 to receive high rate stimulation first), 2 subjects randomized to first receive low rate stimulation were withdrawn prior to stimulation due to difficulties implanting the device. Thus, 18 out of 20 enrolled subjects (9 from each group) started their first intervention.
Groups:
- Low Rate Followed By High Rate: The Precision Plus spinal cord stimulation screening trial leads were temporarily implanted by the investigator. Subjects in this group first received 2 Hz stimulation for 3-4 days, followed by 1200 Hz stimulation for another 3-4 days.
- High Rate Followed By Low Rate: The Precision Plus spinal cord stimulation screening trial leads were temporarily implanted by the investigator. Subjects in this group first received 1200 Hz stimulation for 3-4 days, followed by 2 Hz stimulation for another 3-4 days.
Period: First Intervention (3-4 Days)
Arm/Group | Low Rate Followed By High Rate | High Rate Followed By Low Rate
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Washout (1 Hour)
Arm/Group | Low Rate Followed By High Rate | High Rate Followed By Low Rate
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Second Intervention (3-4 Days)
Arm/Group | Low Rate Followed By High Rate | High Rate Followed By Low Rate
Started | 9 | 9
Completed | 8 | 9
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline measurements were taken for all enrolled subjects (n = 20), but 2 subjects randomized to first receive low rate stimulation withdrew prior to stimulation. Thus, 11 subjects in that group had baseline measurements, but only 9 of them received stimulation.
Groups:
- Low Rate Followed By High Rate: Precision Plus Spinal Cord Stimulation system: The Precision Plus spinal cord stimulation screening trial leads were temporarily implanted by the investigator. Subjects in this group first received 2 Hz stimulation for 3-4 days, followed by 1200 Hz stimulation for another 3-4 days.
- High Rate Followed By Low Rate: Precision Plus Spinal Cord Stimulation system: The Precision Plus spinal cord stimulation screening trial leads were temporarily implanted by the investigator. Subjects in this group first received 1200 Hz stimulation for 3-4 days, followed by 2 Hz stimulation for another 3-4 days.
- Total: Total of all reporting groups
Arm/Group | Low Rate Followed By High Rate | High Rate Followed By Low Rate | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (10.57) | 49.4 (9.49) | 56.5 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 9 | 8 | 17
  Hispanic or Latino | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Back Pain Intensity
Description: Back pain intensity was measured on a 0-10 numerical rating scale (0="no pain", 10="worst pain imaginable") at baseline and following low rate and high rate stimulation. This outcome measure compared the change in intensity from baseline between low rate and high rate stimulation.
Time Frame: For this measure, outcome was assessed at baseline, the end of the first intervention (3 or 4 days post-implantation, depending on the subject), and the end of the second intervention (6 or 8 days post-implantation, depending on the subject).
Measure: Mean (Standard Deviation); unit: Percent Change From Baseline
Groups:
- Low Rate Subperception Precision SCS Trial Therapy: Stimulation was given at a rate of 2 Hz as either a first or second intervention.
- High Rate Subperception Precision SCS Trial Therapy: Stimulation was given at a rate of 1200 Hz as either a first or second intervention.
Arm/Group | Low Rate Subperception Precision SCS Trial Therapy | High Rate Subperception Precision SCS Trial Therapy
Number analyzed (Participants) | 18 | 17
Percent Change From Baseline | 20.9 (31.6) | 25.6 (38.1)
Statistical Analysis 1: Comparison: Low Rate Subperception Precision SCS Trial Therapy vs High Rate Subperception Precision SCS Trial Therapy; Test type: Superiority or Other; p = 0.74, ANOVA; Period effect p=0.11

ADVERSE EVENTS:
Time Frame: 7-9 days
Description: Trial lead insertion was on Day 0, followed by 2 study periods lasting 3-4 days each. Though 18 subjects started stimulation, 20 subjects enrolled and had procedures performed. Two subjects withdrew after attempted lead insertion but before stimulation. Thus, the "At Risk" population during trial lead insertion is reported as 20, not 18.
Groups:
- Trial Lead Insertion: All subjects (n = 20) underwent a lead insertion procedure prior to beginning Period 1 of stimulation. Two of these subjects did not proceed to Period 1 due to insertion difficulties.
- Low Frequency Stimulation: Stimulation was given at 2 Hz.
- High Frequency Stimulation: Stimulation was given at 1200 Hz.
Arm/Group | Trial Lead Insertion | Low Frequency Stimulation | High Frequency Stimulation
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 1/18 | 5/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trial Lead Insertion (N=20) | Low Frequency Stimulation (N=18) | High Frequency Stimulation (N=18)
Administration Site Condition (Device Stimulation Issues) (General disorders) | 0 (0) | 1 | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No